CLINICAL TRIAL: NCT03680079
Title: Group Education Program for High-risk Youth With Poorly-controlled Type 1 Diabetes
Brief Title: High Risk Youth With Poorly-controlled Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201807091
Record Dates: First submitted 2018-09-10; First posted 2018-09-21 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: social media; noncompliance; youth; group education
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Compliance

STUDY DESIGN:
Intervention Model Description: The intervention being studied is a group education program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth with type 1 diabetes (Other): A group of 16 teens (ages 13-18) with poorly -controlled type 1 diabetes will be recruited to participate in this study.
  Interventions: Other: Group education sessions

INTERVENTIONS:
Other: Group education sessions — Peer support and interaction both in-person during group education sessions and online via social media platforms
  Other Names: Social media peer support

SUMMARY:
This study aims to implement a group education curriculum integrated with social media participation to provide peer support and interactive education sessions with the goal of improving glycemic control in disadvantaged youth with poorly-controlled type 1 diabetes.

DETAILED DESCRIPTION:
It has been well established through The Diabetes Control and Complications Trial (DCCT) and its follow-up Epidemiology of Diabetes Interventions and Complications (EDIC) studies that achieving lower hemoglobin A1c (HbA1c) levels are associated with the delay and prevention of long-term complications of T1DM (1, 2). Management of T1DM involves adherence to a complex, labor-intensive regimen of subcutaneous insulin treatment, close glucose monitoring, accurate calculation of carbohydrate intake, and adjustment of dosing and dietary regimen to account for physical activity.

Recent technological advances including insulin pumps with auto-insulin-adjusting features along with continuous glucose monitoring systems have allowed for individuals with T1DM to achieve tighter diabetes control. However, despite these advances in glucose monitoring and insulin delivery systems, the majority of children and adolescents fail to optimize their diabetes control and are unable to achieve these targets.

Several studies have shown that adolescents in poor diabetes control are more likely to come from a racial minority background, have lower annual household income, and be publicly insured. In addition, these patients are also more likely to have missed medical appointments and have less stable home environments. Thus, increased efforts and innovative programs are needed to overcome additional barriers faced by youth with T1DM from disadvantaged backgrounds with the goal of improving the delivery of diabetes care for our most vulnerable, at-risk youth population.

The objective of this pilot and feasibility project is to implement a clinic-based group education program targeting teens with poorly controlled diabetes, focusing on peer group interaction and education combined with social media support to increase engagement and promote behavioral change to improve glycemic control.

This study utilizes 1) group education sessions (6 total sessions over the course of 9 months), 2) online social media group forums, 3) questionnaires to assess self-care habits in diabetes management and quality of life, and 4) surveys to assess this program.

Patients will be included in closed, private Facebook, Snapchat, and Instagram groups where members can communicate with each other and where biweekly updates, reminders, and messages of encouragement relevant to the previous topic covered at group sessions can be sent to the group. Online group forums will be moderated by a staff member to ensure that message content is appropriate and to avoid misinformation or questionable patient-to-patient medical advice.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages 13-18 (at the time of consent) with diagnosis of T1DM
2. HbA1c >9% and/or episode of DKA within the past year (other than at diagnosis)
3. Residence in a zip code associated with lower socioeconomic status (SES)
4. Possession of a device capable of accessing online social media platforms

Exclusion criteria:

1. Non-English speaking
2. Diagnosed with a developmental or psychological condition that would prevent assumption of self-care responsibilities

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 months
  Measure of glycemic control

SECONDARY OUTCOMES:
Diabetes self-management skills | 9 months
  Questionnaire (Self-Care Inventory--Revised Edition) to assess self-management skills prior to and after participation in this study.
  The questionnaire is a validated measure of perceptions of adherence to recommended diabetes self-care behaviors. There are a total of 15 questions, each with a number answer from a scale of "1" to "5". The lowest possible total score is 15, representing poor compliance with diabetes self-management skills, and the highest possible total score would be 75.
Improved quality of life | 9 months
  Peds QL Diabetes Module Version 3.0, Teen Report. This is a validated questionnaire to assess quality of life related to diabetes, this will be filled out at the start and after participation in this study. The questionnaire consists of 28 questions with answers from a scale of "0" to "4" with higher scores representing lower quality of life.
Number of hospital admissions for DKA | 12 months
  Measure of severe diabetes episodes
Depression screening | 9 months
  The PHQ-2 depression questionnaire is a validated 2 question screen for depression.
  Each question has an answer scale from "0" to "3". A score of 3 or more (highest score would be 6) is a positive screen for depression.
  This questionnaire will be given to participants at the start and after participation in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kim, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DCCT/EDIC research group. Effect of intensive diabetes treatment on albuminuria in type 1 diabetes: long-term follow-up of the Diabetes Control and Complications Trial and Epidemiology of Diabetes Interventions and Complications study. Lancet Diabetes Endocrinol. 2014 Oct;2(10):793-800. doi: 10.1016/S2213-8587(14)70155-X. Epub 2014 Jul 17. PMID 25043685
- [Background] Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Study Research Group. Intensive Diabetes Treatment and Cardiovascular Outcomes in Type 1 Diabetes: The DCCT/EDIC Study 30-Year Follow-up. Diabetes Care. 2016 May;39(5):686-93. doi: 10.2337/dc15-1990. Epub 2016 Feb 9. PMID 26861924
- [Background] Campbell MS, Schatz DA, Chen V, Wong JC, Steck A, Tamborlane WV, Smith J, Beck RW, Cengiz E, Laffel LM, Miller KM, Haller MJ; T1D Exchange Clinic Network. A contrast between children and adolescents with excellent and poor control: the T1D Exchange clinic registry experience. Pediatr Diabetes. 2014 Mar;15(2):110-7. doi: 10.1111/pedi.12067. Epub 2013 Aug 19. PMID 23957219
- [Background] Khanolkar AR, Amin R, Taylor-Robinson D, Viner RM, Warner JT, Stephenson T. Young people with Type 1 diabetes of non-white ethnicity and lower socio-economic status have poorer glycaemic control in England and Wales. Diabet Med. 2016 Nov;33(11):1508-1515. doi: 10.1111/dme.13079. Epub 2016 Feb 23. PMID 26802317
- [Background] Fortin K, Pries E, Kwon S. Missed Medical Appointments and Disease Control in Children With Type 1 Diabetes. J Pediatr Health Care. 2016 Jul-Aug;30(4):381-9. doi: 10.1016/j.pedhc.2015.09.012. Epub 2015 Nov 7. PMID 26559135